CLINICAL TRIAL: NCT02867579
Title: Pregnancy Denial and Attachment
Acronym: Denial-attach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PN11015
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy

ARMS (2):
- women with denial pregnancy (Other): women with denial pregnancy
  Interventions: Behavioral: evaluation of the child quality attachment ("Strange situation")
- women without denial pregnancy (Other): women without denial pregnancy
  Interventions: Behavioral: evaluation of the child quality attachment ("Strange situation")

INTERVENTIONS:
Behavioral: evaluation of the child quality attachment ("Strange situation")

SUMMARY:
Described in the 1970's, pregnancy denial occurs as the un-consciousness of being pregnant for several months or throughout the entire period. Body transformations are most of the time not clearly noticeable. The prevalence of this symptom could represent 2 or 3 births over 1000. The definition of pregnancy denial remains unclear due to the different nosological classifications used. There is no international consensus. Encountered terminologies are different from on author to another: pregnancy denial, pregnancy negation. The difficulties to define properly pregnancy denial accurately reflect the clinic heterogeneity of our patients when practicing on a daily basis. As a result, it is difficult to find predictive factors: any women of childbearing age, regardless her age, parity or social professional category, can be subjected to pregnancy denial. Several publications report observations of case of denial of pregnancy, few retrospective studies were realized, only two studies were interested in the future of the child, and no prospective study was interested in the future of the relation mother - child. The denial of pregnancy questions the maternal psychic functioning. No link between psychiatric disorder and denial of pregnancy was until then established. Our various clinical meetings, with mothers having presented a denial of pregnancy and reporting a difficult personal history with many breaks and events susceptibly traumatic, brought us to emit the following hypothesis: an insecure attachment of the mother would participate or at least would facilitate in the construction of a denial of pregnancy. These mothers would have a difficult access, even impossible for the infantile experiences, the essential experiences in the psychic reorganizations of the pregnancy that prepare the woman to accept her new functions of mother. The investigators hypothesize that the attachment and the development of the child, as well as interactions mothers-babies are disturbed when the woman presents a denial of pregnancy.

The research will compare the maternal functioning in both constituted groups (group denial of pregnancy versus groups control), by estimating the type of maternal attachment, without omitting to look for a possible psychiatric pathology, and a personality problem at the mother.

From the questioning on the psychodynamic considerations of the denial of pregnancy, and also on the future of the dyade mother-baby, the investigators construct a national program of clinical research called "Attachment and pregnancy denial", with the participation of 13 centers in France. This research is a prospective cohort examination with main objectives: study the impact of the denial of pregnancy on the pattern of attachment of the child, on the interactions of dyads mother-child and on the early development of the child with a 20-month follow-up. It's a multicenter case-control study with 13 centers (Reims, Strasbourg, Besançon, Nancy, Toulouse, Amiens, Troyes, Toulon, Limoges, Ile-de-France, Lille, Bordeaux, Paris 18ème), to find the maternal risks factors associated to pregnancy denial (secondary objectives).

The main objectives of this study are: (i) studying the relationship between pregnancy denial and the attachment pattern of the child; (ii) studying the relationship between pregnancy denial and the early interactions of mother-infant dyads; (iii) studying the relationship between pregnancy denial and the early development of the child.

The secondary objectives of this study are: (i) studying the relationship between the duration period from the pregnancy announcement to the delivery and the early development of a child, including the attachment pattern of a child, the early interactions of mother-infant dyads, (ii) looking for the risk factors associated to pregnancy denial, including the type of attachment, the existence of a personality disorders and/or a psychiatric pathology

DETAILED DESCRIPTION:
The follow-up of the cases and the witnesses will be identically and carried out according to the following process: First visit (post-delivery, at the maternity): reception of the informed consent, collection of demographic data (age, marital status, level of education, financial resources), social data (life form, socio-economic data of the child father, developmental data of the child siblings) and medical records (gestation and parity, pregnancy records, medical surgical and psychiatric history). During the first examination: evaluation by perceived social support self-questionnaire (QSSP) and MNI (Psychiatric disorders Axis I). Second visit (during the mandatory post-natal consultation, 6 to 8 weeks after delivery): Evaluation by self-questionnaires of depression (BDI and EPDS), maternal anxiety (STAI), and personality disorders (screening IPDE) and evaluation of maternal attachment pattern (AAN). Third visit (when the child is 6 months old, at the mother's home): video recording to evaluate the interactions during a meal (CIB), self-questionnaires of the child temperament (QT6) and maternal depression (EPDS), evaluation of the child development (Denver scale), evaluation of a relational retreat behaviour of the child (ADBB), semi-structured interview for the personality disorders (IPDE). Fourth visit (when the child is 12 months old, at the mother's home): maternal self-questionnaires (BDI, STAI, QSSP, EPDS), video recording to evaluate the interactions during a meal (CIB), evaluation of the child development (Denver scale), evaluation of a relational retreat behaviour of the child (ADBB). Fifth visit (when the child is 18 months old, in a room equipped with video recording): evaluation of the child quality attachment ("Strange situation"), evaluation of the child development (Denver scale). Sixth visit (when the child is 20 months old, at the mother home): open conversation with the mother.

The total duration of participation of a patient is of 20 months.

Will be analysed in this study, the impact of pregnancy denial as well as the duration period from the pregnancy announcement to the delivery on: (i) The attachment pattern of the child, evaluated by the "Strange Situation". A mother and a child are under observation in a laboratory. The observer notes the child reactions during 8 episodes of 3 minutes involving the separations and reunions between the mother and the child, as well as the introduction of a stranger. The situation is observed behind a two-way mirror and recorded in video. This procedure of evaluation of the attachment was organized according to the Mary Ainsworth's works. The coding system of interactive behaviours allows a categorization into 4 attachment patterns: "secure", "anxious-avoidant insecure" "anxious-ambivalent resistant insecure" and "disorganized/disoriented and insecure" (Regrouped into two categories: "Secure" and "Insecure"). (ii) The quality of early interactions between the mother and the child evaluated by the Coding Interactive Behaviour (CIB - Feldman) (10), the CIB includes 42 items (21 concerning the mother, 16 concerning the child and 5 concerning the dyad). Each item is evaluated on a 5 points scale. The scale consists of 2 segmentations of 15 minutes interactions: one episode of game and one episode of feeding. (iii) The infant's temperament characteristics evaluated by the QT6 (Infant Characteristics Questionnaire, Bates), specific questions will be asked to parents about the "difficult" temperament of the child. The filling lasts approximately 10 minutes, the questionnaire account 26 questions. It was validated in France with 794 mothers of old children from 6 to 9 months, by the team of the Dr B. Larroque. (iiii) The child's development evaluated by the Denver scale (DSST - Denver Developmental Screening Test), the child is accessed in different areas such as gross motor skills, language, fine motor skills, and social contact, and by the ADBB scale. This scale includes 8 items concerning facial expression, eye contact, body activity, self-simulation gestures and fingers activities, level of vocal expression, liveliness of a response to stimulation, ability to connect with someone else and attractiveness.

Research for factors potentially associated to the occurrence of a denial of pregnancy: (i) Pattern of mother's attachment evaluated by the AAN (Adult Attachment Narratives), it allows studying the representations of the attachment at the adult through the analysis of 4 narratives (2 referring in the relations over adults, and 2 in the relations mother - child) built by the subject. He is asked to use 12 words by narrative presented in writing by the examiner (these words establishing the weft of the history). These narratives are blind recorded and analyzed by professionals trained and validated in the scale, every narrative receives a note of 1 in 7 reflecting the secure base of the script in connection with the pattern of attachment of the subject. The average obtained in these 4 narratives estimates the security of attachment of the subject and allows the categorization in 2 groups notes = 3: pattern of attachment insecure, notes > 3 pattern of attachment secure). The interview lasts approximately 1/2 the hour. The entire interview is transcribed verbatim to allow the quotation. (ii) Mother's personality evaluated with the IPDE (International Personality Disorders Examination) is a semi-structured diagnosis interview allowing the evaluation of personality disorders described in the CIM 10. It contains 67 items. The criteria of personality are grouped in six domains: work, personal, interpersonal relations, affects, apprehension of the reality and the control of the impulses. The administration of the instrument varies between 60 and 90 minutes. (iii) Mother's psychiatric trouble assesses with the MINI (Mini International Neurospychiatric Interview) is a structured diagnostic maintenance, exploring the main psychiatric disorders of the axis I of the CIM 10. It contains 120 questions and is divided into 16 modules, each corresponding in a diagnosis category: A. Major depressive disorder, B. Dysthymia, C. Suicidal risk, D. Mania (hypomania) episode, E. Panic disorder, F. Agoraphobia, G. Social phobia, F. Obsessive-compulsive disorder, I. Post-traumatic stress disorder, J. Alcohol (dependence / abuse), K. Drugs (dependence / abuse), L. Psychotic disorders, M. Anorexia nervosa, N. Bulimia nervosa, O. Generalized anxiety disorder, and P. Antisocial personality Disorder. For each of the disorders(confusions), two in four questions-filters are presented at the beginning of every module, allowing the screening. The signing of the MINI is brief, on average 19 minutes. The MINI was simultaneously developed in French and in English.

To neutralize the identified biases, we also assess maternal comorbidities: (i) Postnatal depression screened with the EPDS (Edinburgh Post-natal Depression Scale), a self-questionnaire of screening of the postnatal depression. EPDS is a quick self-questionnaire used in Anglo-Saxon countries since its elaboration by John Cox in 1987, validated by a number of studies, translated and validated for France by Nicole Guedeney in 1995. The formulation is simple and its easy use. We consider a known postnatal depression when the score is upper or equal to 11. (ii) Maternal anxiety evaluated with the scale STAI (Trait Anxiety Inventory) form Y, Trait Anxiety Inventory of Spielberger. The inventory of trait anxiety is intended to estimate on one hand the trait anxiety and on the other hand the state anxiety through 20 items, which concern only the psychological and not somatic aspects of the anxiety. The Y version was developed to eliminate items more bound to the depression. "State Trait Inventory Anxiety" is both very used in the practice and in the clinical research. It includes different scales to estimate the state (STAI form Y-A) and the trait (STAI form Y-B). Each scale includes 20 proposals, the scale E to estimate what the subjects feel at the moment, the scale T to seize what the subjects feel generally. The STAI is intended for the auto-administration. He can be individually performed or in a group. The time of signing is about 10 minutes to fill in both scales. Every answer to a proposal of the questionnaire corresponds to a score from 1 to 4: - 1 indicating the lowest degree of anxiety, - 4 the strongest degree. French translation and validation by Scweitzer MB. (iii) Maternal depression evaluated with the scale BDI (Beck Depression Inventory), it gives a quantitative estimation of the intensity of the depressive feelings. It includes 21 items of symptoms and attitudes, which describe a specific behavior of the depression, increased from 0 to 3 by a series of 4 statements reflecting the severity degree of the symptom. Scale translated and validated in French by P. Bourque and D. Beaudette, on 1982. (iiii) Maternal social support estimated by the Perceived Social Support Questionnaire (QSSP), a self-assessment that estimates the availability and the satisfaction with the social support received. The authors were inspired by the theory of the attachment of Bowlby, by associating the notion of social support with fundamental needs: need for proximity with the mother, then need for a relation favoured with others significant. Thus this scale allows estimating the type of received support, the sources of this support, number of people who get it (or availability) and the perceived quality (or satisfaction). This tool also informs about the nature of the social support perceived by the person. Translated in French by Bruchon-Schweitzer, Rascle, Sarason.

ELIGIBILITY:
Inclusion Criteria:

* women with pregnancy denial defined by a pregnancy announcement after 20 weeks of gestation and a lack of objectives perception of the pregnancy by the woman and delivery in the previous week
* women without pregnancy denial and delivery in the previous week
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* For women with pregnancy announcement after 20 weeks of gestation : No follow-up of the pregnancy due to geographical reason, social reason (no insurance coverage) and administrative reason: Mothers facing family conflicts: multiparous or marital conflicts; Mothers facing social difficulties: unemployment, hidden pregnancy to the employer.
* women with intellectual disabilities,
* women with acute or chronic psychotic disorders,
* women who doesn't speak properly French,
* born to an unidentified mother,
* women who received a PMA treatment during pregnancy.
* newborn with life threatening prognostic or with an organic malformation and/or genetic - abnormality observed before leaving maternity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
child quality attachment | 18 months
  evaluation of the child quality attachment using "Strange situation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Auer J, Barbe C, Sutter AL, Dallay D, Vulliez L, Riethmuller D, Gubler V, Verlomme V, Saad-Saint-Gilles S, Miton A, Tessier E, Parant O, Le Foll J, Bourgeois-Moine A, Viaux S, Dommergues M, Apter G, Belaisch-Allart J, Danion A, Nisand I, Graesslin O, Novo A, Eutrope J, Rolland AC. Pregnancy denial and early infant development: a case-control observational prospective study. BMC Psychol. 2019 Apr 11;7(1):22. doi: 10.1186/s40359-019-0290-3. PMID 30971319
- [Result] Delong H, Eutrope J, Thierry A, Sutter-Dallay AL, Vulliez L, Gubler V, Saad Saint-Gilles S, Tessier E, Le Foll J, Viaux S, Apter G, Danion A, Auer J, Rolland AC; Pregnancy Denial Study Group. Pregnancy denial: a complex symptom with life context as a trigger? A prospective case-control study. BJOG. 2022 Feb;129(3):485-492. doi: 10.1111/1471-0528.16853. Epub 2021 Aug 19. PMID 34324258